CLINICAL TRIAL: NCT02256371
Title: Efficacy of 2 Psycho-physical Methods in the Treatment of Neuropathic Pain: a Randomized Controlled Monocentric Study
Brief Title: Randomized Controlled Study of the Efficacy of Hypnosis Versus Relaxation and Control in Neuropathic Pain
Acronym: PSYCNEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130604
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Hypnosis; Relaxation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hypnotic analgesia (Experimental): Hypnosis sessions:
  Hypnosis will consist of 45 minutes hypnosis session with a trained hypnotherapist
  Interventions: Behavioral: Hypnosis sessions
- Relaxation (Experimental): Relaxation group:
  Relaxation will be conducted in 45 minutes sessions with a trained psychotherapist.
  Interventions: Behavioral: Relaxation group
- Routine care (No Intervention): The patients will receive their usual pain treatments throughout the study

INTERVENTIONS:
Behavioral: Hypnosis sessions — 1 session per week during 8 weeks
  Arms: Hypnotic analgesia
Behavioral: Relaxation group — 1 relaxation session per week during 8 weeks
  Arms: Relaxation

SUMMARY:
A randomized double-blind controlled two centers study. The primary objective of this study will be to show a superiority of hypnosis over relaxation on pain intensity in patients with neuropathic pain.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* to show a superiority of hypnosis and relaxation over control group on neuropathic pain.
* to show a lasting effect of treatment on neuropathic pain one week after the end of treatment.
* to evaluate the clinical predictors of response to hypnosis (nature of neuropathic symptoms, severity of anxiety and depressive symptoms, pain catastrophizing, coping strategies, emotional regulation, response to the first session, positive or negative emotional reaction at the end of hypnosis sessions).
* to evaluate the effect of hypnosis at long-term (1, 3 and 6 months after the end of treatment).
* to evaluate the effect of hypnosis on emotional processes.
* to compare hypnosis to relaxation on short-term effects on pain,
* to evaluate the quality of life and the impact of pain on daily life: sleep, mood, anxiety symptoms, analgesics consumption , neuropathic symptoms, affective component of pain and pain catastrophizing.

  35 patients will be enrolled in each arm, to obtain 105 in total (3 arms). Total duration for each patient: 8 months.

ELIGIBILITY:
Inclusion Criteria:

* peripheral or central neuropathic pain, probable or definite
* Diagnostic questionnaire score DN4 ≥ 4/10
* Chronic Pain with an average of pain intensity greater than or equal to 4/10 (digital scale)
* Presence of daily or almost daily pain (i.e. at least 4 days per week)
* Patient with pre-existing pain for > 6 months
* Patient > 18 and < 60 years old
* Patient with a stable analgesic treatment since 15 days before inclusion
* Patient able to participate to the trial during 33 weeks
* Patient having a health insurance
* Written informed consent signed by the patient.

Exclusion Criteria:

* Prior treatment with hypnosis
* Currently under active psychotherapy (Cognitive-Behavior Therapy, psychoanalysis)
* Work accident or litigation
* Drugs abuse or Psychoactive Substance Abuse (DSM-IV)
* Neuropathic pain associated with progressive disease (MS, HIV, cancer ...)
* Major depression with ongoing disability or psychosis (DSM IV)
* Intermittent pain
* Patient with pre-existing pain for < 6 months
* Other more severe pain than the pain justifying inclusion
* Subject unable to understand the trial information provided in the informed consent document
* Subject under curators or guardianship
* Severe Handicap or amputation
* Participation to another study in the same period
* Deafness
* Cognitive disorders (dementia, Mild Cognitive Impairment, inability to understand the questionnaires)
* For patients of the control arm: Treatment by hypnosis and / or relaxation, transcranial magnetic stimulation, or invasive treatments (surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Weekly mean pain intensity in patients diaries | 9 week
  The pain intensity score will be recorded daily by each patient on a self-assessment diary using a scale of 0 to 10. The record will begin from the first session of hypnosis or relaxation to the last session (S1 to S9).

SECONDARY OUTCOMES:
Pain intensity measured at the end of each visit and 3 and 6 months after the end of the treatment | 8 months
  Pain intensity measured at the end of each hypnosis or relaxation session and 3 and 6 months after the end of the treatment
Evaluation of the feeling of comfort and relaxation | 9 weeks
  At the end of each hypnosis or relaxation session, with a scale from 0 to 10.
Affective components of pain | 8 months
  At the end of each visit and 3 and 6 months after the end of the treatment
Emotional processes and Alexithymia | 8 months
Neuropathic symptoms (NPSI) | 8 months
Interference with pain (Brief Pain Inventory) | 8 months
Quality of life assessment | 8 months
Depression and anxiety | 8 months
Emotional distress caused by pain | 8 months
Pain catastrophizing | 9 months
Pain relief | 8 months
Delay of onset of analgesic effects | 8 weeks
Percentage of responders | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD, PhD, Principal Investigator — Groupe Hospitalier Ambroise Paré
Locations (1):
- Centre d'évaluation et de traitement de la douleur, Hôpital Ambroise Paré, Boulogne-Billancourt, Hauts-de-Seine, France